CLINICAL TRIAL: NCT04040829
Title: Cognitive Remediation and Supported Education in Psychotic Disorders: a Randomized Controlled Trial on the Efficacy and the Best Predictors of Academic Functioning
Brief Title: Cognitive Remediation and Supported Education in Psychotic Disorders
Acronym: REUSSIR
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: A feasibility study will be conducted to assess the online administration of the cognitive remediation program CIRCuiTS.
Sponsor: Centre de Recherche de l'Institut Universitaire en Santé Mentale de Québec (Other)
Collaborators: Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Caroline Cellard, Associate professor, Centre de Recherche de l'Institut Universitaire en Santé Mentale de Québec
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MP-13-2019-1538, NSM (MP)
Record Dates: First submitted 2019-07-29; First posted 2019-08-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Psychotic Disorders
Keywords: Cognitive remediation therapy; Supported education; Academic functioning; Schizophrenia; Cognition; Photovoice; Mixed qualitative and quantitative methodology
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This study is a two arm single blind randomized trial comparing Cognitive remediation therapy + Supported education + Treatment as usual with Supported Education + Treatment as usual alone
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blind to treatment allocation, but patients, cognitive remediation therapists and supported education specialists will not be blind. We will ask participants to not disclose their group allocation to the assessor. Furthermore, each patient will be assessed by a different assessor for each time point (T0, T1, T2, T3) to ensure blindness.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SE + TAU (Active Comparator): Supported education (SE) includes a variety of services ranging from orientation, study strategies or homework help. This intervention is personalized to the need of each patient in terms of services and frequency. Previous to this randomized controlled trial, we conducted interviews with each site that will provide SE. In these interviews, we explored the fidelity of their services to the Individual Placement and Support adapted to education. Information regarding the dosage of SE (frequency, length of session, type of support) will be collected and used as covariates for each participant since intensity treatment can impact outcomes.
  Treatment as usual (TAU) consists of medication and routine contact with the clinical team. Patients will continue to receive their standard treatment, but we will collect information regarding the type of medication, the dosage, and all other relevant information and use it as covariate in our analyses.
  Interventions: Behavioral: Supported education (SE); Other: Treatment as usual (TAU)
- CR + SE + TAU (Experimental): Cognitive remediation therapy (CR) will be conducted using CIRCuiTS, a computerized program designed to improve cognition (attention, memory, executive functioning) and metacognitive skills. CIRCuiTS has an integrated focus on the transfer of cognitive skills to daily living, using real-world goals and homework to facilitate in vivo use of new strategies, as well as a formulation-based approach, which takes into account the impact of cognitive strengths and difficulties with daily living skills. Each session includes about 4-8 tasks targeting a range of cognitive problems, which become more ecologically valid as the program progresses. The rate of delivery for CIRCuiTS will be two to three sessions per week, for a maximum of 40 sessions. The therapy will be provided entirely online with a therapist, using the platform Zoom.
  This arm will include our active control condition : supported education (SE) as well as Treatment as usual (TAU) as previously described.
  Interventions: Behavioral: Cognitive remediation therapy (CR); Behavioral: Supported education (SE); Other: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Cognitive remediation therapy (CR) — Cognitive remediation therapy is a behavioral intervention that aims to improve cognition. This intervention has the goal to produce long-term improvements in cognition as well as to generalize these improvements in daily functioning.
  Arms: CR + SE + TAU
Behavioral: Supported education (SE) — Supported education (SE) is a behavioral intervention that aims to help people return to school and/or succeed in school. SE offers a wide range of services that are personalized to the needs of each patients.
Other: Treatment as usual (TAU) — Treatment as usual (TAU) consists of medication and routine contact with the clinical team.

SUMMARY:
This trial aims to assess the added value of cognitive remediation therapy to supported education intervention in young adults with a psychotic disorder. The objectives of this study are threefold: The first objective is to evaluate the efficacy of supported education and cognitive remediation therapy for young adults with psychotic disorders in terms of academic outcome (primary outcome) and cognitive, neurobiological, and psychological outcomes (secondary outcomes). The second objective is to explore mechanisms of change in academic outcomes using a multidimensional approach (cognitive, psychological and biological characteristics) in youth with psychotic disorders. The third objective is to investigate the patients' perspectives regarding their appreciation of the supported education programs.

Academic outcomes, cognitive performance as well as psychological and genetic variables will collected at baseline (T0). Participants will then be randomized either to the experimental condition (Cognitive remediation + Supported education + Treatment as usual) or the control condition (Supported education + Treatment as usual) for three months. Directly after the end of treatment (T1) and three months following the end of treatment (T2), the same measures as baseline will be repeated. One year post-treatment (T3), a last assessment will be conducted for academic outcomes.To assess qualitative experience of patients enrolled in supported education, a subsample of the randomized controlled trial will be recruited to participate in a photovoice activity.

DETAILED DESCRIPTION:
Psychotic disorders often occur during late adolescence and early adulthood. Cognitive deficits are among the most debilitating features of these disorders and have important impacts on academic functioning. Youth with psychotic disorders are more likely drop-out or to struggle completing high school and entering postsecondary education. Supported education programs (SE) help people with mental illness succeed in school by providing various services. However, these programs do not target cognitive deficits. Cognitive remediation therapy (CR) is an evidence-based cost-effective treatment to improve cognitive deficits. CR leads to significant improvements in cognition, symptoms and functioning, and improvements are even larger when combined with psychiatric rehabilitation interventions, such as supported employment. However, little attention has been paid to SE. Combining CR and SE is an integrative approach that could have a positive effect on academic functioning in youth with psychotic disorders.

This trial aims to assess the added value of cognitive remediation therapy to supported education intervention in young adults with a psychotic disorder. The objectives of this study are threefold: The first objective is to evaluate the efficacy of supported education and cognitive remediation therapy for young adults with psychotic disorders in terms of academic outcome (primary outcome) and cognitive, neurobiological, and psychological outcomes (secondary outcomes). The second objective is to explore mechanisms of change in academic outcomes using a multidimensional approach (cognitive, psychological and biological characteristics) in youth with psychotic disorders. The third objective is to investigate the patients' perspectives regarding their appreciation of the supported education programs.

Participants will be assessed at baseline (T0) using a multidimensional approach including academic outcomes as well as cognitive, psychological and genetic measures. Participants will then be randomized to the experimental condition (Cognitive remediation + Supported education + Treatment as usual) or the control condition (Supported education + Treatment as usual) for three months. The cognitive remediation program that will be used is CIRCuiTS (Computerised Interactive Remediation of Cognition Training for Schizophrenia). Directly after the end of treatment (T1) and three months following the end of treatment (T2), the same measures as baseline will be repeated. One year post-treatment (T3), a last assessment will be conducted for academic outcomes.

To assess qualitative experience of patients enrolled in supported education, a subsample of the randomized controlled trial will be recruited to participate in a photovoice activity. Photovoice is a participatory research approach that enables vulnerable people to act as co-researchers by identifying and representing their personal experience through photography or video. This approach notably includes a life-book approach in which participants will document their experience through photos they will take and other images they can find on the web or any other media, which will be paired with a narrative interview focusing on documenting their significant experiences going through the intervention.

ELIGIBILITY:
Inclusion Criteria:

* aged from 16 to 35 years
* diagnosis of a psychotic disorder as confirmed by a psychiatrist
* currently enrolled or in the process of enrollment in a supported education program
* performance more than one standard deviation below the normative mean of the participant age and sex normative group in one of the following cognitive functions: episodic memory, working memory, attention, speed of processing or executive function

Exclusion Criteria:

* evidence of an organic cause of cognitive difficulties
* plans to change medication during the study
* receiving concurrently another type of therapy (e.g. Cognitive Behavioral Therapy (CBT), etc.)

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline on the First-Episode Social Functioning Scale (School subscale) | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The FESFS assesses different aspect of functioning including social functioning, productive activities and instrumental activities of daily living. Each question is rated on a Likert scale ranging from 1=Totally disagree to 4= Completely agree. The School subscale assesses the ability to meet deadlines, punctuality and school performance.
Mean change from baseline on the First-Episode Social Functioning Scale (School subscale) | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The FESFS assesses different aspect of functioning including social functioning, productive activities and instrumental activities of daily living. Each question is rated on a Likert scale ranging from 1=Totally disagree to 4= Completely agree. The School subscale assesses the ability to meet deadlines, punctuality and school performance.
Mean change from baseline on the First-Episode Social Functioning Scale (School subscale) | Baseline (T0; moment of enrollment in the study) to 1-year post-treatment (T3; one year following the end of the intervention)
  The FESFS assesses different aspect of functioning including social functioning, productive activities and instrumental activities of daily living. Each question is rated on a Likert scale ranging from 1=Totally disagree to 4= Completely agree. The School subscale assesses the ability to meet deadlines, punctuality and school performance.
Mean change from baseline on the First-Episode Social Functioning Scale (Relationships and social activities at school subscale) | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The FESFS assesses different aspect of functioning including social functioning, productive activities and instrumental activities of daily living. Each question is rated on a Likert scale ranging from 1=Totally disagree to 4= Completely agree. Relationships and social activities at school subscale assesses relationships with professors and students as well as participation in class.
Mean change from baseline on the First-Episode Social Functioning Scale (Relationships and social activities at school subscale) | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The FESFS assesses different aspect of functioning including social functioning, productive activities and instrumental activities of daily living. Each question is rated on a Likert scale ranging from 1=Totally disagree to 4= Completely agree. Relationships and social activities at school subscale assesses relationships with professors and students as well as participation in class.
Mean change from baseline on the First-Episode Social Functioning Scale (Relationships and social activities at school subscale) | Baseline (T0; moment of enrollment in the study) to 1-year post-treatment (T3; one year following the end of the intervention)
  The FESFS assesses different aspect of functioning including social functioning, productive activities and instrumental activities of daily living. Each question is rated on a Likert scale ranging from 1=Totally disagree to 4= Completely agree. Relationships and social activities at school subscale assesses relationships with professors and students as well as participation in class.
Mean change from baseline on the Rubric tool | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The Rubric tool assesses six domains of academic functioning, namely contributions, attitude, preparedness, focus on the task, professionalism and effort, and a composite score from those six scales. Based on the rating of several questions, a mean score of each domain, as well as a total score, will be obtained using a Likert scale that ranges from 1 (lowest the student can achieve) to 4 (highest the student can achieve).
Mean change from baseline on the Rubric tool | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The Rubric tool assesses six domains of academic functioning, namely contributions, attitude, preparedness, focus on the task, professionalism and effort, and a composite score from those six scales. Based on the rating of several questions, a mean score of each domain, as well as a total score, will be obtained using a Likert scale that ranges from 1 (lowest the student can achieve) to 4 (highest the student can achieve).
Mean change from baseline on the Rubric tool | Baseline (T0; moment of enrollment in the study) to 1-year post-treatment (T3; one year following the end of the intervention)
  The Rubric tool assesses six domains of academic functioning, namely contributions, attitude, preparedness, focus on the task, professionalism and effort, and a composite score from those six scales. Based on the rating of several questions, a mean score of each domain, as well as a total score, will be obtained using a Likert scale that ranges from 1 (lowest the student can achieve) to 4 (highest the student can achieve).

SECONDARY OUTCOMES:
Raw score change from baseline on the California verbal learning test-II (CVLT-II) (delayed recall). | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The CVLT-II assesses verbal episodic memory. The test includes the learning of a list of words, followed by an immediate and a delayed recall.
Raw score change from baseline on the California verbal learning test-II (CVLT-II) (delayed recall). | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The CVLT-II assesses verbal episodic memory. The test includes the learning of a list of words, followed by an immediate and a delayed recall.
Raw score change from baseline on the Rey Complex Figure test (delayed recall). | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The Rey complex figure test assesses visual episodic memory. The test includes the copy of a complex figure, followed by an immediate and a delayed recall.
Raw score change from baseline on the Rey Complex Figure test (delayed recall). | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The Rey complex figure test assesses visual episodic memory. The test includes the copy of a complex figure, followed by an immediate and a delayed recall.
Raw score change from baseline on the digit span subtest backward of the Wechsler Adult Intelligence Scale-IV (WAIS-IV) | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The digit span subtest backward assesses verbal working memory. A series of number are read to the participant. The participant has to recall the numbers backward.
Raw score change from baseline on the digit span subtest backward of the Wechsler Adult Intelligence Scale-IV (WAIS-IV) | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The digit span subtest backward assesses verbal working memory. A series of number are read to the participant. The participant has to recall the numbers backward.
Raw score change from baseline on the coding subtest of the Wechsler Adult Intelligence Scale-IV (WAIS-IV) | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The coding subtest assesses speed of processing. The participant has to match as many numbers as possible with symbols based on a key.
Raw score change from baseline on the coding subtest of the Wechsler Adult Intelligence Scale-IV (WAIS-IV) | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The coding subtest assesses speed of processing. The participant has to match as many numbers as possible with symbols based on a key.
Raw score change from baseline on the spatial span subtest backward of the Wechsler Memory Scale | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The spatial span subtest backward assesses visual working memory. A board with blocks are presented to the participant. The assessor point series of blocks and the participant has to point the blocks backward.
Raw score change from baseline on the spatial span subtest backward of the Wechsler Memory Scale | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The spatial span subtest backward assesses visual working memory. A board with blocks are presented to the participant. The assessor point series of blocks and the participant has to point the blocks backward.
Raw score change from baseline on the Hit Reaction Time Block Change (HRT-BC) of the Continuous Performance Test-3 (CPT-3) | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The HRT-BC assesses sustained attention. Letters appear on a computer screen and the participant has to press the space bar as fast as possible, except when the letter is an "X". The HRT-BC reflects the reaction time between the six conditions of the CPT-3. In each condition, the letters are presented at a different rate. A higher HRT-BC score indicates a decrease of efficiency in information processing, which suggest difficulties in sustained attention.
Raw score change from baseline on the Hit Reaction Time Block Change (HRT-BC) of the Continuous Performance Test-3 (CPT-3) | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The HRT-BC assesses sustained attention. Letters appear on a computer screen and the participant has to press the space bar as fast as possible, except when the letter is an "X". The HRT-BC reflects the reaction time between the six conditions of the CPT-3. In each condition, the letters are presented at a different rate. A higher HRT-BC score indicates a decrease of efficiency in information processing, which suggest difficulties in sustained attention.
Raw score change from baseline on the fourth condition of the Trail Making Test (Delis-Kaplan Executive Function System; D-KEFS) | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The fourth condition of the Trail Making Test assesses cognitive flexibility. Letters and numbers are presented on a page.The participants has to connect these letters in alphabetical order and the numbers in numerical order while alternating between the numbers and letters
Raw score change from baseline on the fourth condition of the Trail Making Test (Delis-Kaplan Executive Function System; D-KEFS) | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The fourth condition of the Trail Making Test assesses cognitive flexibility. Letters and numbers are presented on a page.The participants has to connect these letters in alphabetical order and the numbers in numerical order while alternating between the numbers and letters
Raw score change from baseline on the third condition of the color-word interference (Delis-Kaplan Executive Function System; D-KEFS) | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The third condition of the color-word interference assesses inhibition. Name of color written in a different color of ink are presented to the participant. The participant has to name the color of the ink for each word as fast as possible.
Raw score change from baseline on the third condition of the color-word interference (Delis-Kaplan Executive Function System; D-KEFS) | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The third condition of the color-word interference assesses inhibition. Name of color written in a different color of ink are presented to the participant. The participant has to name the color of the ink for each word as fast as possible.
Raw score change from baseline on the verbal fluency subtest (first condition) (Delis-Kaplan Executive Function System; D-KEFS) | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The first condition of the verbal fluency subtest assesses phonemic fluency. The participant has to name as many word as possible in one minute that start by a given letter.
Raw score change from baseline on the verbal fluency subtest (first condition) (Delis-Kaplan Executive Function System; D-KEFS) | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The first condition of the verbal fluency subtest assesses phonemic fluency. The participant has to name as many word as possible in one minute that start by a given letter.
Raw score change from baseline on the Tower of London (total item completed with the minimum movement) | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The Tower of London assesses planning and organization. For this test, the assessor produces different models on his board using three beads (green, blue and red). The participant has to replicate the model using as few moves as possible.
Raw score change from baseline on the Tower of London (total item completed with the minimum movement) | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The Tower of London assesses planning and organization. For this test, the assessor produces different models on his board using three beads (green, blue and red). The participant has to replicate the model using as few moves as possible.
Raw score change from baseline on the Matrix subtest of the Wechsler Adult Intelligence Scale-IV (WAIS-IV) | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The Matrix reasoning subtest assesses perceptual reasoning. Series of complex patterns are presented to the participant. The participant has to choose the logical end to each pattern.
Raw score change from baseline on the Matrix subtest of the Wechsler Adult Intelligence Scale-IV (WAIS-IV) | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The Matrix reasoning subtest assesses perceptual reasoning. Series of complex patterns are presented to the participant. The participant has to choose the logical end to each pattern.
Raw score change from baseline on the Combined Stories test | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The Combined stories test assesses theory of mind. Short stories are presented to the participant and questions regarding the mental states of the characters are asked.
Raw score change from baseline on the Combined Stories test | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The Combined stories test assesses theory of mind. Short stories are presented to the participant and questions regarding the mental states of the characters are asked.
Raw score change from baseline on the Social Knowledge test | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The Social Knowledge test assess social perception. Situations of daily life are presented to the participant. The participant is asked to state the emotion that would be felt by most people in that situation.
Raw score change from baseline on the Social Knowledge test | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The Social Knowledge test assess social perception. Situations of daily life are presented to the participant. The participant is asked to state the emotion that would be felt by most people in that situation.
Raw score change from baseline on the Penn Emotion Recognition task | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The Penn Emotion Recognition task assesses emotion recognition. Faces expressing emotions are presented on a computer screen. The participant has to determine the emotion expressed by the character among the seven choices.
Raw score change from baseline on the Penn Emotion Recognition task | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The Penn Emotion Recognition task assesses emotion recognition. Faces expressing emotions are presented on a computer screen. The participant has to determine the emotion expressed by the character among the seven choices.
Raw score change from baseline on the Échelle de Répercussion Fonctionnelle | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The Échelle de Répercussion Fonctionnelle assesses functional impact of cognitive deficits in daily living using a semi-structured interview. The severity of the functional impact is rated on a Likert scale from 1= no impact to 7=important impact.
Raw score change from baseline on the Échelle de Répercussion Fonctionnelle | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The Échelle de Répercussion Fonctionnelle assesses functional impact of cognitive deficits in daily living using a semi-structured interview. The severity of the functional impact is rated on a Likert scale from 1= no impact to 7=important impact.
Raw score change from baseline on the Positive And Negative Syndrome Scale (PANSS) | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The PANSS is a semi-structured interview that assess clinical symptoms of psychotic disorder, including positive symptoms, negative symptoms and general psychopathology.
Raw score change from baseline on the Positive And Negative Syndrome Scale (PANSS) | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The PANSS is a semi-structured interview that assess clinical symptoms of psychotic disorder, including positive symptoms, negative symptoms and general psychopathology.
Raw score change from baseline on the Self-Esteem Rating Scale (SERS) | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The SERS assesses self-esteem. The questionnaire includes 20 questions rated on a Likert scale from 1=Never to 7=Always
Raw score change from baseline on the Self-Esteem Rating Scale (SERS) | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The SERS assesses self-esteem. The questionnaire includes 20 questions rated on a Likert scale from 1=Never to 7=Always
Raw score change from baseline on the Subjective Scale to Investigate Cognition in Schizophrenia (SSTICS) | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The SSTICS assesses metacognitive knowledge, i.e., participant' perceptions of his cognitive abilities. The questionnaire includes 21 questions rated on a Likert scale ranging from 0=Never to 4=very often.
Raw score change from baseline on the Subjective Scale to Investigate Cognition in Schizophrenia (SSTICS) | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The SSTICS assesses metacognitive knowledge, i.e., participant' perceptions of his cognitive abilities. The questionnaire includes 21 questions rated on a Likert scale ranging from 0=Never to 4=very often.
Raw score change from baseline on the First-Episode Social Functioning Scale (FESFS) | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The FESFS assesses different aspect of functioning including social functioning, productive activities and instrumental activities of daily living. Each question is rated on a Likert scale ranging from 1=Totally disagree to 4= Completely agree
Raw score change from baseline on the First-Episode Social Functioning Scale (FESFS) | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The FESFS assesses different aspect of functioning including social functioning, productive activities and instrumental activities of daily living. Each question is rated on a Likert scale ranging from 1=Totally disagree to 4= Completely agree
Raw score change from baseline on the Childhood Trauma Questionnaire (CTQ) | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  The CTQ assesses adverse events experienced during childhood and adolescence. The CTQ includes 70 items rated on a Likert scale ranging from 1=Never true to 5=very often true
Raw score change from baseline on the Childhood Trauma Questionnaire (CTQ) | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  The CTQ assesses adverse events experienced during childhood and adolescence. The CTQ includes 70 items rated on a Likert scale ranging from 1=Never true to 5=very often true
Presence or absence of a genetic variant (Met66Met) of the Brain-derived neurotrophic factor (BDNF) gene (Val66Met) at baseline | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  Presence or absence of a genetic variant (Met66Met) of the BDNF gene (Val66Met).
Presence or absence of a genetic variant (Met66Met) of the Brain-derived neurotrophic factor (BDNF) gene (Val66Met) at baseline | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  Presence or absence of a genetic variant (Met66Met) of the BDNF gene (Val66Met).
Presence or absence of the Val158Met polymorphism on the Catechol-O-Methyltransferase (COMT) gene | Baseline (T0; moment of enrollment in the study) to Post-treatment (T1; directly after the 3-months period of intervention)
  Single nucleotide polymorphisms (SNP) in the 3' end of the COMT gene and the Val158Met polymorphism
Presence or absence of the Val158Met polymorphism on the Catechol-O-Methyltransferase (COMT) gene | Baseline (T0; moment of enrollment in the study) to 3-months post-treatment (T2; three months following the end of the intervention)
  Single nucleotide polymorphisms (SNP) in the 3' end of the COMT gene and the Val158Met polymorphism

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Cellard, Ph.D, Principal Investigator — Centre de Recherche de l'Institut Universitaire en Santé Mentale de Québec; Tania Lecomte, Ph.D, Principal Investigator — Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal; Marc Corbière, Ph.D, Principal Investigator — Université du Québec a Montréal
Locations (3):
- Canada (3):
  - Centre de recherche de l'Institut universitaire en santé mentale de Montréal, Montreal, Quebec
  - Centre hospitalier universitaire de Montréal, Montreal, Quebec
  - Centre de recherche CERVO, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Achim AM, Ouellet R, Roy MA, Jackson PL. Mentalizing in first-episode psychosis. Psychiatry Res. 2012 Apr 30;196(2-3):207-13. doi: 10.1016/j.psychres.2011.10.011. Epub 2012 Feb 28. PMID 22377576
- [Background] Bell M, Bryson G, Greig T, Corcoran C, Wexler BE. Neurocognitive enhancement therapy with work therapy: effects on neuropsychological test performance. Arch Gen Psychiatry. 2001 Aug;58(8):763-8. doi: 10.1001/archpsyc.58.8.763. PMID 11483142
- [Background] Bond GR, Drake RE, Becker DR. Generalizability of the Individual Placement and Support (IPS) model of supported employment outside the US. World Psychiatry. 2012 Feb;11(1):32-9. doi: 10.1016/j.wpsyc.2012.01.005. PMID 22295007
- [Background] Bosia M, Bechi M, Marino E, Anselmetti S, Poletti S, Cocchi F, Smeraldi E, Cavallaro R. Influence of catechol-O-methyltransferase Val158Met polymorphism on neuropsychological and functional outcomes of classical rehabilitation and cognitive remediation in schizophrenia. Neurosci Lett. 2007 May 7;417(3):271-4. doi: 10.1016/j.neulet.2007.02.076. Epub 2007 Mar 2. PMID 17383818
- [Background] Bosia M, Zanoletti A, Spangaro M, Buonocore M, Bechi M, Cocchi F, Pirovano A, Lorenzi C, Bramanti P, Smeraldi E, Cavallaro R. Factors affecting cognitive remediation response in schizophrenia: the role of COMT gene and antipsychotic treatment. Psychiatry Res. 2014 Jun 30;217(1-2):9-14. doi: 10.1016/j.psychres.2014.02.015. Epub 2014 Feb 19. PMID 24656901
- [Background] Carmona VR, Gomez-Benito J, Huedo-Medina TB, Rojo JE. Employment outcomes for people with schizophrenia spectrum disorder: A meta-analysis of randomized controlled trials. Int J Occup Med Environ Health. 2017 May 8;30(3):345-366. doi: 10.13075/ijomeh.1896.01074. Epub 2017 Apr 26. PMID 28481370
- [Background] Cellard C, Reeder C, Paradis-Giroux AA, Roy MA, Gilbert E, Ivers H, Bouchard RH, Maziade M, Wykes T. A feasibility study of a new computerised cognitive remediation for young adults with schizophrenia. Neuropsychol Rehabil. 2016;26(3):321-44. doi: 10.1080/09602011.2015.1019891. Epub 2015 Mar 10. PMID 25753694
- [Background] Corbiere M, Bond GR, Goldner EM, Ptasinski T. Brief reports: the fidelity of supported employment implementation in Canada and the United States. Psychiatr Serv. 2005 Nov;56(11):1444-7. doi: 10.1176/appi.ps.56.11.1444. PMID 16282266
- [Background] Cutler DM, Lleras-Muney A. Education and health: evaluating theories and evidence (No. w12352). National bureau of economic research, 2006
- [Background] Davidson L. Living outside mental illness: qualitative studies of recovery in schizophrenia, University Press, New York, 2003
- [Background] Day JC, Newburger EC. The Big Payoff: Educational Attainment and Synthetic Estimates of Work-Life Earnings. Special Studies. Current Population Reports, 2002
- [Background] Delis DC, Kramer J, Kaplan E, Ober, B. CVLT-II. San Antonio, TX: The Psychological Corporation, 2000
- [Background] Diaz-Asper CM, Goldberg TE, Kolachana BS, Straub RE, Egan MF, Weinberger DR. Genetic variation in catechol-O-methyltransferase: effects on working memory in schizophrenic patients, their siblings, and healthy controls. Biol Psychiatry. 2008 Jan 1;63(1):72-9. doi: 10.1016/j.biopsych.2007.03.031. Epub 2007 Aug 20. PMID 17707347
- [Background] Fett AK, Viechtbauer W, Dominguez MD, Penn DL, van Os J, Krabbendam L. The relationship between neurocognition and social cognition with functional outcomes in schizophrenia: a meta-analysis. Neurosci Biobehav Rev. 2011 Jan;35(3):573-88. doi: 10.1016/j.neubiorev.2010.07.001. Epub 2010 Jul 8. PMID 20620163
- [Background] Fisher M, Mellon SH, Wolkowitz O, Vinogradov S. Neuroscience-informed Auditory Training in Schizophrenia: A Final Report of the Effects on Cognition and Serum Brain-Derived Neurotrophic Factor. Schizophr Res Cogn. 2016 Mar 1;3:1-7. doi: 10.1016/j.scog.2015.10.006. PMID 26705516
- [Background] Goulding SM, Chien VH, Compton MT. Prevalence and correlates of school drop-out prior to initial treatment of nonaffective psychosis: further evidence suggesting a need for supported education. Schizophr Res. 2010 Feb;116(2-3):228-33. doi: 10.1016/j.schres.2009.09.006. Epub 2009 Sep 24. PMID 19783405
- [Background] Greco V, Lambert HC, Park M. Being visible: PhotoVoice as assessment for children in a school-based psychiatric setting. Scand J Occup Ther. 2017 May;24(3):222-232. doi: 10.1080/11038128.2016.1234642. Epub 2016 Sep 26. PMID 27665933
- [Background] Harvey PD, Green MF, Keefe RS, Velligan DI. Cognitive functioning in schizophrenia: a consensus statement on its role in the definition and evaluation of effective treatments for the illness. J Clin Psychiatry. 2004 Mar;65(3):361-72. PMID 15096076
- [Background] Ikegame T, Bundo M, Murata Y, Kasai K, Kato T, Iwamoto K. DNA methylation of the BDNF gene and its relevance to psychiatric disorders. J Hum Genet. 2013 Jul;58(7):434-8. doi: 10.1038/jhg.2013.65. Epub 2013 Jun 6. PMID 23739121
- [Background] Jemal A, Thun MJ, Ward EE, Henley SJ, Cokkinides VE, Murray TE. Mortality from leading causes by education and race in the United States, 2001. Am J Prev Med. 2008 Jan;34(1):1-8. doi: 10.1016/j.amepre.2007.09.017. PMID 18083444
- [Background] Karpova NN. Role of BDNF epigenetics in activity-dependent neuronal plasticity. Neuropharmacology. 2014 Jan;76 Pt C:709-18. doi: 10.1016/j.neuropharm.2013.04.002. Epub 2013 Apr 12. PMID 23587647
- [Background] Kohler CG, Turner TH, Bilker WB, Brensinger CM, Siegel SJ, Kanes SJ, Gur RE, Gur RC. Facial emotion recognition in schizophrenia: intensity effects and error pattern. Am J Psychiatry. 2003 Oct;160(10):1768-74. doi: 10.1176/appi.ajp.160.10.1768. PMID 14514489
- [Background] Kidd SA, Kaur J, Virdee G, George TP, McKenzie K, Herman Y. Cognitive remediation for individuals with psychosis in a supported education setting: a randomized controlled trial. Schizophr Res. 2014 Aug;157(1-3):90-8. doi: 10.1016/j.schres.2014.05.007. Epub 2014 Jun 2. PMID 24893903
- [Background] Killackey E, Allott K, Woodhead G, Connor S, Dragon S, Ring J. Individual placement and support, supported education in young people with mental illness: an exploratory feasibility study. Early Interv Psychiatry. 2017 Dec;11(6):526-531. doi: 10.1111/eip.12344. Epub 2016 Apr 28. PMID 27121481
- [Background] Nuechterlein KH, Subotnik KL, Ventura J, Turner LR, Gitlin MJ, Gretchen-Doorly D, Becker DR, Drake RE, Wallace CJ, Liberman RP. Enhancing return to work or school after a first episode of schizophrenia: the UCLA RCT of Individual Placement and Support and Workplace Fundamentals Module training. Psychol Med. 2020 Jan;50(1):20-28. doi: 10.1017/S0033291718003860. Epub 2019 Jan 4. PMID 30606273
- [Background] Lecomte T, Corbiere M, Ehmann T, Addington J, Abdel-Baki A, Macewan B. Development and preliminary validation of the First Episode Social Functioning Scale for early psychosis. Psychiatry Res. 2014 May 30;216(3):412-7. doi: 10.1016/j.psychres.2014.01.044. Epub 2014 Feb 5. PMID 24613006
- [Background] Lecomte T, Corbiere M, Laisne F. Investigating self-esteem in individuals with schizophrenia: relevance of the Self-Esteem Rating Scale-Short Form. Psychiatry Res. 2006 Jun 30;143(1):99-108. doi: 10.1016/j.psychres.2005.08.019. Epub 2006 May 24. PMID 16725210
- [Background] McGurk SR, Mueser KT, Feldman K, Wolfe R, Pascaris A. Cognitive training for supported employment: 2-3 year outcomes of a randomized controlled trial. Am J Psychiatry. 2007 Mar;164(3):437-41. doi: 10.1176/ajp.2007.164.3.437. PMID 17329468
- [Background] McGurk SR, Mueser KT, DeRosa TJ, Wolfe R. Work, recovery, and comorbidity in schizophrenia: a randomized controlled trial of cognitive remediation. Schizophr Bull. 2009 Mar;35(2):319-35. doi: 10.1093/schbul/sbn182. Epub 2009 Mar 5. PMID 19269925
- [Background] Medalia A, Saperstein AM, Hansen MC, Lee S. Personalised treatment for cognitive dysfunction in individuals with schizophrenia spectrum disorders. Neuropsychol Rehabil. 2018 Jun;28(4):602-613. doi: 10.1080/09602011.2016.1189341. Epub 2016 May 24. PMID 27219068
- [Background] Meyers JE, Meyers KR. Rey Complex Figure Test and recognition trial professional manual. Psychological Assessment Resources, 1995
- [Background] Nuechterlein KH, Subotnik KL, Green MF, Ventura J, Asarnow RF, Gitlin MJ, Yee CM, Gretchen-Doorly D, Mintz J. Neurocognitive predictors of work outcome in recent-onset schizophrenia. Schizophr Bull. 2011 Sep;37 Suppl 2(Suppl 2):S33-40. doi: 10.1093/schbul/sbr084. PMID 21860045
- [Background] Nykiforuk CI, Vallianatos H, Nieuwendyk LM. Photovoice as a Method for Revealing Community Perceptions of the Built and Social Environment. Int J Qual Methods. 2011 Jan 1;10(2):103-124. doi: 10.1177/160940691101000201. PMID 27390573
- [Background] Panizzutti R, Hamilton SP, Vinogradov S. Genetic correlate of cognitive training response in schizophrenia. Neuropharmacology. 2013 Jan;64(1):264-7. doi: 10.1016/j.neuropharm.2012.07.048. Epub 2012 Aug 7. PMID 22992330
- [Background] Pieramico V, Esposito R, Sensi F, Cilli F, Mantini D, Mattei PA, Frazzini V, Ciavardelli D, Gatta V, Ferretti A, Romani GL, Sensi SL. Combination training in aging individuals modifies functional connectivity and cognition, and is potentially affected by dopamine-related genes. PLoS One. 2012;7(8):e43901. doi: 10.1371/journal.pone.0043901. Epub 2012 Aug 28. PMID 22937122
- [Background] Reeder C, Harris V, Pickles A, Patel A, Cella M, Wykes T. Does change in cognitive function predict change in costs of care for people with a schizophrenia diagnosis following cognitive remediation therapy? Schizophr Bull. 2014 Nov;40(6):1472-81. doi: 10.1093/schbul/sbu046. Epub 2014 Mar 28. PMID 24682210
- [Background] Reeder C, Huddy V, Cella M, Taylor R, Greenwood K, Landau S, Wykes T. A new generation computerised metacognitive cognitive remediation programme for schizophrenia (CIRCuiTS): a randomised controlled trial. Psychol Med. 2017 Nov;47(15):2720-2730. doi: 10.1017/S0033291717001234. Epub 2017 Sep 4. PMID 28866988
- [Background] Reeder C, Wykes T. Computerised Interactive Remediation of Cognition - Interactive Training for Schizophrenia (CIRCUITS). London: Kings College London, 2010
- [Background] Stip E, Caron J, Renaud S, Pampoulova T, Lecomte Y. Exploring cognitive complaints in schizophrenia: the subjective scale to investigate cognition in schizophrenia. Compr Psychiatry. 2003 Jul-Aug;44(4):331-40. doi: 10.1016/S0010-440X(03)00086-5. PMID 12923712
- [Background] Suijkerbuijk YB, Schaafsma FG, van Mechelen JC, Ojajarvi A, Corbiere M, Anema JR. Interventions for obtaining and maintaining employment in adults with severe mental illness, a network meta-analysis. Cochrane Database Syst Rev. 2017 Sep 12;9(9):CD011867. doi: 10.1002/14651858.CD011867.pub2. PMID 28898402
- [Background] Thibaudeau E, Cellard C, Reeder C, Wykes T, Ivers H, Maziade M, Lavoie MA, Pothier W, Achim AM. Improving Theory of Mind in Schizophrenia by Targeting Cognition and Metacognition with Computerized Cognitive Remediation: A Multiple Case Study. Schizophr Res Treatment. 2017;2017:7203871. doi: 10.1155/2017/7203871. Epub 2017 Jan 26. PMID 28246557
- [Background] Tsang HW, Leung AY, Chung RC, Bell M, Cheung WM. Review on vocational predictors: a systematic review of predictors of vocational outcomes among individuals with schizophrenia: an update since 1998. Aust N Z J Psychiatry. 2010 Jun;44(6):495-504. doi: 10.3109/00048671003785716. PMID 20482409
- [Background] Vauth R, Corrigan PW, Clauss M, Dietl M, Dreher-Rudolph M, Stieglitz RD, Vater R. Cognitive strategies versus self-management skills as adjunct to vocational rehabilitation. Schizophr Bull. 2005 Jan;31(1):55-66. doi: 10.1093/schbul/sbi013. Epub 2005 Feb 16. PMID 15888425
- [Background] Wang C, Burris MA. Photovoice: concept, methodology, and use for participatory needs assessment. Health Educ Behav. 1997 Jun;24(3):369-87. doi: 10.1177/109019819702400309. PMID 9158980
- [Background] Wechsler D. Wechsler intelligence scale for children (4th ed.). San Antonio, TX: The Psychological Corporation, 2008
- [Background] Wykes T, Huddy V, Cellard C, McGurk SR, Czobor P. A meta-analysis of cognitive remediation for schizophrenia: methodology and effect sizes. Am J Psychiatry. 2011 May;168(5):472-85. doi: 10.1176/appi.ajp.2010.10060855. Epub 2011 Mar 15. PMID 21406461